CLINICAL TRIAL: NCT04278287
Title: A Phase I/II Study of Chemoradiotherapy Using Albumin-Bound Paclitaxel and Cisplatin in Unresectable Esophageal Squamous Cell Carcinomas Based on Nutritional Risk Screening Score (NRS2002)
Brief Title: Chemoradiotherapy in Unresectable Esophageal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XIN WANG, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/325-2109
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer; Chemoradiotherapy; Albumin-bound Paxlitaxel; Unresectable Malignant Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Cisplatin; Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Albumin-Bound Paclitaxel and Cisplatin based chemoradiotherapy (Experimental): Chemoradiotherapy arm receives intensity-modulated radiation therapy, volume modulated arc therapy or tomotherapy concurrently with albumin-bound paclitaxel and cisplatin (weekly intravenous infusion in 5-6 weeks).
  Interventions: Radiation: Radiotherapy; Drug: Albumin-Bound Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiotherapy — 59.92Gy and 2.14Gy in 28 fractions to PGTV and 50.4Gy and 1.8Gy in 28 fractions 5 days every week in 5.5 weeks.
Drug: Albumin-Bound Paclitaxel — 100mg/d weekly,repeatedly on the first day,by intravenous infusion in 5-6 weeks.
  Other Names: Nab-Paclitaxel
Drug: Cisplatin — 25mg/m2 weekly,by intravenous infusion in 5-6 weeks.
  Other Names: platinum

SUMMARY:
This phase I/II clinical study is designed to evaluate the 1 year local tumor control rate of chemoradiotherapy using albumin-bound paclitaxel and cisplatin in unresectable esophageal squamous cell carcinomas based on Nutritional Risk Screening NRS2002.

DETAILED DESCRIPTION:
This Phase I/II clinical study is meticulously designed to assess the one-year local tumor control rate of a chemoradiotherapy regimen that combines albumin-bound paclitaxel and cisplatin in patients with unresectable esophageal squamous cell carcinoma (ESCC). The selection of participants is guided by the Nutritional Risk Screening (NRS2002) tool, which ensures that nutritional risk factors are adequately considered and managed throughout the study.

The trial will enroll patients diagnosed with unresectable ESCC, a condition where surgical intervention is not feasible due to the tumor's location, size, or patient comorbidities. Participants will undergo a thorough nutritional assessment using the NRS2002 criteria, which evaluates factors such as weight loss, body mass index, dietary intake, and severity of disease to determine their nutritional risk score. This screening is crucial as it helps identify patients who may benefit from nutritional interventions, which could potentially improve their overall response to the treatment and quality of life.

Once enrolled, patients will receive a combination chemoradiotherapy of albumin-bound paclitaxel and cisplatin. Albumin-bound paclitaxel is chosen for its ability to improve the delivery and efficacy of paclitaxel, a chemotherapy drug, by enhancing its solubility and distribution within the body. Cisplatin, a platinum-based chemotherapy agent, is included due to its well-established efficacy in treating various cancers, including esophageal cancer. This combination aims to maximize tumor reduction while managing potential side effects.

The primary endpoint of the study is to determine the local tumor control rate at one year, which refers to the percentage of patients whose tumors have not progressed or recurred within the treated area during this period. Secondary endpoints include overall survival, progression-free survival, and assessment of treatment-related toxicity. Additionally, the study will monitor changes in patients' nutritional status and quality of life, aiming to provide comprehensive insights into the efficacy and safety of this chemoradiotherapy regimen.

Regular follow-ups and imaging studies, such as CT scans or PET scans, will be conducted to evaluate the tumor response and detect any signs of progression. Blood tests and other laboratory assessments will be performed periodically to monitor patients' overall health and manage any adverse effects promptly. The data collected from this study will contribute valuable information to the ongoing efforts to improve treatment outcomes for patients with unresectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18~75 years
* Pathologically or cytologically proven unresectable esophageal squamous cell carcinomas in patients staged as T3N1M0-1b and T4N0-1M0-1b(AJCC 6th TNM staging,M1b limited to clavicular or celiac lymph node metastasis)
* Primary treatment performed in Cancer Hospital, Chinese Academy of Medical Sciences
* ECOG PS score: 0~1
* NRS2002 score <3
* Estimated survival time ≥3 months
* Normal organ and marrow function as defined below:

Hemoglobin: greater than or equal to 100g/L ;Leukocytes: greater than or equal to 4,000 G/L; Neutrophil: greater than or equal to 2,000 G/L; Platelets: greater than or equal to 100,000/mm3 ; Creatinine: less than or equal to 1.5 times the upper limit or CCR greater than or equal to 60 ml/min; AST/ALT: less than or equal to 2.5 times the upper limit; Total bilirubin: less than or equal to 1.5 times the upper limit; INR: less than or equal to 1.5 times the upper limit; APTT: less than or equal to 1.5 times the upper limit; PT: less than or equal to 1.5 times the upper limit

* Informed consent

Exclusion Criteria:

* With any distant metastasis out of regional lymphatic drainage or in liver, lung, bone, CNS, etc
* Patients with other cancer history in 5 years except cervical carcinoma in situ and non-malignant melanoma skin cancer
* Existing active infection such as active tuberculosis and hepatitis
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of allergic reactions attributed to paclitaxel, albumin or cisplatin
* Participation in other clinical trials currently or within 4 weeks of selection
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 1 year from the start of treatment to tumor recurrence
  Control rate of primary esophageal cancer and metastatic lymph nodes within irradiation fields

SECONDARY OUTCOMES:
Number of participants with acute toxicities | 10 week, from the start of treatment to 1 month after chemoradiotherapy
  Acute toxicities are evaluated by NCI-CTC version 5.0
Objective response rate | 5.5 week
  Objective Response Rate are evaluated by RECIST 1.1
Disease Free Survival | 1 year, 2 year
  The time from treatment to progression or death
Progression Free Survival | 1 year, 2 year
  The time from treatment to progression or death
Overall Survival | 1 year, 2 year
  The time from treatment to death from any cause
Radiomics analysis | 5.5 week
  Radiomics analysis for tumor response and survival prediction with pre- and post-chemoradiotherapy based on MRI and CT simulation
ctDNA analysis | 4 week, 2 month, 1 year, 2 year
  ctDNA analysis to monitor therapeutic efficacy including tumor response and survival outcome

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (5):
- China (5):
  - Department 4th of Radiation Oncology, Anyang Cancer Hospital, Anyang, Henan
  - Hunan Cancer Hospital, the Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - Department of Radiation oncology, Jiangsu Cancer Hospital/Jiangsu Institute of Cancer Research/The affiliated Cancer Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Department of Radiation oncology, Jiangsu Province Hospital/The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Department of Radiation Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing